CLINICAL TRIAL: NCT03448354
Title: Comparative Effectiveness of HIPEC Following Interval Debulking Surgery in Patients With Advanced-stage Ovarian Cancer Undergoing Neoadjuvant Chemotherapy: Multicenter, Prospective, Cohort Study
Brief Title: Comparative Effectiveness of HIPEC Following Interval Debulking Surgery in Patients With Advanced-stage Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Suk-Joon Chang, Director, Division of Gynecologic Oncology; Professor, Department of Obstetrics and Gynecology, Ajou University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-OBS-17-324
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Cancer
Keywords: HIPEC; Interval debulking surgery
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness of HIPEC following interval debulking surgery in patients with advanced-stage ovarian cancer undergoing neoadjuvant chemotherapy: Multicenter, prospective, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC-IDS-HIPEC (Experimental): Under the clinicians' decision, HIPEC procedures will be performed at the time of IDS.
  Interventions: Procedure: HIPEC
- NAC-IDS (No Intervention): Under the clinicians' decision, HIPEC procedures will not be performed at the time of IDS.

INTERVENTIONS:
Procedure: HIPEC — HIPEC(paclitaxel 175mg/m2, 90min; open or closed technique) after IDS . IDS is recommended within 4 weeks after the 3rd NAC cycle. HIPEC procedure is allowed only in case of residual disease less than 5mm.
  Arms: NAC-IDS-HIPEC

SUMMARY:
Ovarian cancer is a lethal malignancy and reported as a fifth leading cause of death in all age in the developed country. Most of the ovarian cancer patients are diagnosed at advanced stages due to an inadequate screening tool and a lack of clinical symptoms. Optimal cytoreductive surgery with no gross residual disease followed platinum-based adjuvant chemotherapy has been the most effective therapeutic strategy in the treatment of advanced ovarian cancer. However, the optimal surgical procedure is not always possible, especially in patients with extensive disease or women with poor performance status. Neoadjuvant chemotherapy(NAC) followed interval debulking surgery (IDS) is an alternative therapeutic option for these patients. There is growing interest in the use of HIPEC (hyperthermic intraperitoneal chemotherapy) for ovarian cancer, and early data on HIPEC as a component of front-line therapy of advanced ovarian cancer are encouraging. However, intraperitoneal chemotherapy is not actively used in the treatment of ovarian cancer due to the catheter-related complications or inconvenience. The aim of this study is to evaluate the effectiveness and safety of HIPEC after interval debulking surgery in advanced ovarian cancer patients.

DETAILED DESCRIPTION:
GOG 172 trial showed a dramatic improvement of overall survival in patients with stage III disease treated with intraperitoneal cisplatin and paclitaxel compared with those with intravenous administration. Currently, prospective cohort study showed a survival benefit of intraperitoneal chemotherapy compared with intravenous chemotherapy. Despite this improvement, intraperitoneal chemotherapy is not widely used as standard therapy owing to the high rate of adverse effects and inconvenience of administering therapy intraperitoneally. Hyperthermic intraperitoneal chemotherapy (HIPEC) is a multi-modal approach with combined intraperitoneal chemotherapy and hyperthermia. It maintains the theoretical benefit of intraperitoneal chemotherapy and reduces most of the adverse events from catheter-related problems with delivery of the chemotherapeutic agent at the end of surgery. In addition, hyperthermia increases the penetration of chemotherapy at the peritoneal surface and chemo-sensitivity. In this trial, we aim to evaluate the efficacy and safety of HIPEC procedures performed after interval debulking surgery in patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. patients histologically diagnosed with EOC (epithelial ovarian cancer), fallopian tubal cancer or primary peritoneal cancer.
2. patients treated with neoadjuvant chemotherapy (NAC) followed by interval debulking surgery due to expected suboptimal residual disease at the time of primary surgery.
3. patients who had diagnostic laparoscopy before NAC and confirmed with tumor burden, Fagotti score ≥8.
4. ECOG performance status (0~2)
5. lab findings Bone marrow function : ANC>1,500/mm3, Platelet >100,000/mm3, Hemoglobin>10.0g/dl Kidney function : creatinine<1.25xUNL Liver function: AST, ALT< x1.5UNL, bilirubin<1.5mg/dl
6. Live expenctancy > 6 month
7. Age > 19 years old

Exclusion Criteria:

1. Patients with treated with primary debulking surgery
2. Patients with double primary cancer ( exception: patients with early breast cancer or endometrial cancer that will not affect the clinical course of ovarian cancer)
3. Patients with pregnant or breast feeding

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 5 years
  From the study enrollment to the disease progression

SECONDARY OUTCOMES:
Response rate | up to 1 years
  rate of patients with partial or complete response (RECIST criteria version 1.1 ) after primary treatment
Overall survival | up to 5 years
  From study enrollment to the patients death
Adverse drug reaction | up to 1 years
  Incidence of grade 3 or 4 drug adverse reaction (NCI CTCAE version 4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Joon Chang, MD, PhD, Principal Investigator — Ajou University
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided